CLINICAL TRIAL: NCT02532673
Title: Impact of Hyperbilirubinemia Among HIV Patients Treated With Atazanavir
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI424-531
Record Dates: First submitted 2015-08-11; First posted 2015-08-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hyperbilirubinemia Cohort: Patients will be included who have evidence of hyperbilirubinemia (laboratory test of grade 2 or greater or > 2 medical claims with an International Classification of Diseases, Ninth Revision, Clinical Modification code of 782.4 or 277.4 in any position) in the first 90 days after initiating Atazanavir therapy.
- Non-hyperbilirubinemia cohort: Patients will be included who have no evidence of hyperbilirubinemia (no laboratory test of grade 2 or greater or any medical claims with an International Classification of Diseases, Ninth Revision, Clinical Modification of 782.4 or 277.4 in any position) in the 12-month follow-up period.

SUMMARY:
The purpose of this study is to determine whether HIV patients on Atazanavir who have Hyperbilirubinemia have different outcomes from those without Hyperbilirubinemia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Human immunodeficiency virus
* Treatment with Atazanavir
* 18 yrs and older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Commercially insured population (single large health plan)
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Atazanavir persistence among treated patients who develop hyperbilirubinemia compared with Atazanavir-treated patients without evidence of hyperbilirubinemia | One year after starting Atazanavir
  Discontinuation rate, defined as proportion of patients having discontinued Atazanavir at 1 year, of HBR vs. non-HBR patients. Persistence, defined as mean days to Atazanavir discontinuation, of HBR vs non-HBR patients. Compliance defined as mean medication-possession ratio of HBR vs non-HBR patients
Atazanavir compliance among treated patients who develop hyperbilirubinemia compared with Atazanavir-treated patients without evidence of hyperbilirubinemia | One year after starting Atazanavir
  Discontinuation rate, defined as proportion of patients having discontinued Atazanavir at 1 year, of HBR vs. non-HBR patients. Persistence, defined as mean days to Atazanavir discontinuation, of HBR vs non-HBR patients. Compliance defined as mean medication-possession ratio of HBR vs non-HBR patients

SECONDARY OUTCOMES:
Healthcare costs for HBR vs non-HBR patients | 1 year
  Health care costs:
  Health care costs will be computed as the combined health plan and patient paid amounts for all claims in the 12-month post-index period. Mean costs will be calculated for total costs, medical costs, pharmacy costs, ambulatory costs, emergency services costs, inpatient costs, and other costs.
  * Costs will be adjusted into 2013 US dollars using the annual medical care component of the Consumer Price Index (CPI) to reflect inflation between 2003 and 2013
Health care resource utilization for HBR vs non-HBR patients | 1 year
  Health care resource utilization:
  Binary indicators and counts of mean number of ambulatory visits (office and outpatient), ER visits, and inpatient admissions over 12 months will be calculated. Total number of inpatient days and mean length of inpatient stay will also will be captured.
Changes (increase, decrease, no change) in the grade of bilirubin laboratory test results during follow-up among Atazanavir-treated patients who develop hyperbilirubinemia | 1 year
  Grade of the bilirubin test result will be captured and defined as follows: Grade 0 = normal; Grade 1 ≥ 1.0 to 1.5 times the upper limit of normal (x ULN), Grade 2 ≥1.5 to 2.5 x ULN; Grade 3 ≥ 2.5 to 5 x ULN; Grade 4 ≥ 5 x ULN
  The upper limit of normal range was used to standardize the laboratory results across different lab systems. Each laboratory vendor provides a normal range for their results. These results were then transformed based on the normal ranges provided. The ranges below were used to categorize the patients:
  =0, if result in normal rage
  =1, if result > 1.0-1.5 times the upper limit of normal (x ULN)
  =2, if result > 1.5-2.5 x ULN
  =3, if result > 2.5-5 x ULN
  =4, if result > 5 x ULN
Rate of Human immunodeficiency virus viral suppression among patients treated with Atazanavir who develop hyperbilirubinemia compared with patients without evidence of hyperbilirubinemia | 1 year
Liver function based on Alanine aminotransferase and Aspartate aminotransferase test results among patients treated with Atazanavir who develop hyperbilirubinemia compared with patients without evidence of hyperbilirubinemia | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx